CLINICAL TRIAL: NCT00708526
Title: Improved Patient Recovery After Anesthesia With Hypercapnia Hyperpnoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Anecare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 26111
Record Dates: First submitted 2008-06-30; First posted 2008-07-02 (Estimated); Results first posted 2011-10-19 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Hypercapnia
Keywords: hypercapnia; hyperpnoea; accelerated recovery
MeSH Terms: conditions — Hypercapnia; Hyperventilation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 Recovery (Experimental): Quick Emergence Device is in place for phase 1 anesthesia recovery
  Interventions: Device: Quick Emergence Device
- Standard of care (Other): Tidal volume and respiratory rate are not changed during phase 1 recovery from anesthesia
  Interventions: Other: standard of care for phase one anesthesia care

INTERVENTIONS:
Other: standard of care for phase one anesthesia care — Patients received intravenous fentanyl at the discretion of the attending anesthesiologist. Anesthesia was induced with a remifentanil infusion, lidocaine, propofol, and rocuronium or succinylcholine at the anesthesiologist's discretion. Maintenance anesthesia was 6% end tidal desflurane with oxygen flows of 2 L/min (though clinicians could deviate from this at their discretion). Clinicians were directed to maintain blood pressure at ±20% of baseline. A baseline remifentanil infusion was used throughout each case, and both remifentanil and fentanyl were titrated at the anesthesiologist's discretion. Ventilation was adjusted to maintain an end tidal carbon dioxide concentration (EtCO2) of 35 mmHg. Ondansetron 4 mg was given prophylactically before the end of surgery.
  Arms: Standard of care
Device: Quick Emergence Device — The Quick Emergence Device is placed between the endotracheal tube and the anesthesia breathing circuit to enable hypercapnia when ventilation is increased. The end-tidal gas sampling line is connected between the device and the endotracheal tube connector. Minute ventilation is doubled and the EtCO2 is elevated to approximately 48 mmHg from the previous maintenance level of 35 mmHg.
  Other Names: QED-100 from Anecare Inc
  Arms: Phase 1 Recovery

SUMMARY:
The proposed study will measure the time from the end of surgery until the time patients meet the discharge criteria from the postoperative anesthesia care unit and the time from the end of surgery until the patients regained cognitive function after anesthesia.

DETAILED DESCRIPTION:
Hypercapnia has been used in conjunction with hyperpnoea to provide a more rapid return of responsiveness after inhaled anesthesia. In our first clinical study with isoflurane we confirmed that the time from turning off the vaporizer to opening of eyes was shortened by an average of 62% when the minute ventilation was elevated and the end tidal carbon dioxide concentration was kept at 52 mmHg rather than 28 mmHg during emergence. In our second study we found that hypercapnia and hyperpnoea accelerated recovery proportionately for sevoflurane and desflurane. The benefits of accelerating subject recovery in the operating room may extend to the entire recovery period if the subject is more alert and easier to care for when they arrive in the post anesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

* adults
* ASA class I-III
* both genders
* scheduled to undergo eye surgery at the Moran Hospital.

Exclusion Criteria:

* a history of renal or hepatic disease,
* chronic alcohol or drug abuse,
* disabling neuropsychiatric disorder,
* hypersensitivity or unusual response to other halogenated anesthetics,
* pulmonary hypertension,
* increased intracranial pressure,
* seizure disorder
* personal/familial history of malignant hyperthermia.
* currently being treated with known hepatic enzyme-inducing drugs (e.g., phenobarbital, dilantin or isoniazid)
* or with drugs known to alter anesthetic requirements (e.g., opiates, clonidine, alpha2 agonists, alcohol, anticonvulsants, antidepressants, barbiturates, benzodiazepines or other tranquilizers).
* intolerance to non-steroidal anti-inflammatories.
* have received general anesthesia within the previous 7 days,
* received any investigational drug within the previous 28 days,
* participated in a previous isoflurane or desflurane study
* Female subjects can be neither pregnant nor breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dwayne Westenskow, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from March 28-August 25, 2008 through the surgery schedule at the Moran Eye Center
Groups:
- Quick Emergence Device (QED): At the end of surgery, the Quick Emergence Device was placed between the endotracheal tube and the anesthesia breathing circuit. Minute ventilation was doubled and the end tidal carbon dioxide concentration (EtCO2) was elevated to approximately 48 mmHg.
- Standard of Care: At the end of surgery, the minute ventilation and EtCO2 remained at normal levels. The Quick Emergence Device was not used.
Period: Wake up After Anesthesia
Arm/Group | Quick Emergence Device (QED) | Standard of Care
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Return of Cognitive Function
Arm/Group | Quick Emergence Device (QED) | Standard of Care
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quick Emergence Device (QED) | Standard of Care | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 43.7 (15.1) | 40.4 (15) | 42.1 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Recovery From Anesthesia
Description: average time in minutes from the time the surgeon finished closing the surgical incision until the time the investigator in the postoperative care unit determined that the patients meet the discharge criteria from the postoperative anesthesia care unit (their vital signs had been stable for at least 30 min, their pain scores were less than the tolerable pain scores, they could sit up without dizziness or nausea, and their Aldrete score was ≥8).
Time Frame: up to 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Quick Emergence Device (QED) | Standard of Care
Number analyzed (Participants) | 11 | 11
minutes | 53.0 (15.2) | 62.9 (28.8)
Statistical Analysis 1: Comparison: Quick Emergence Device (QED) vs Standard of Care; We compared times for discharge criteria after general anesthesia with and without the QED; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; A Bonferroni correction was used

2. Secondary Outcome: Return of Cognitive Function
Description: average time in minutes from the time the surgeon finished closing the surgical incision at the end of surgery until the patients could correctly state their full name, the current year and their day, month and year of birth
Time Frame: up to 30 minutes
Population: number of participants determined by protocol
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Quick Emergence Device (QED) | Standard of Care
Number analyzed (Participants) | 11 | 11
minutes | 10.9 (5.1) | 18.2 (9.7)
Statistical Analysis 1: Comparison: Quick Emergence Device (QED) vs Standard of Care; The effect of the use of hypercapnia and increased ventilation on the time to recovery events was compared using multivariate analysis of variance with the Hotelling's two sample T2.-test and the two-tailed unpaired t-test; individual comparisons were by Bonferroni adjusted two tailed unpaired t-tests. The data was tested for normality before identifying statistical significance; Test type: Superiority or Other; p = 0.039, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Quick Emergence Device (QED) | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes